CLINICAL TRIAL: NCT02840812
Title: Pharmacokinetics Study of Nemonoxacin Malate Capsules in Subjects With Severe Impaired Renal Function
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: XCNN-150830-2
Record Dates: First submitted 2016-07-19; First posted 2016-07-21 (Estimated); Last update posted 2018-04-03 (Actual); Status verified 2018-04

CONDITIONS: Kidney Dysfunction
MeSH Terms: interventions — nemonoxacin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Renal function impaired (Experimental): Subject with Severe Impaired Renal Function. Nemonoxacin Malate Capsules 500mg single dose oral
  Interventions: Drug: Nemonoxacin
- Healthy Subjects (Experimental): Healthy volunteers. Nemonoxacin Malate Capsules 500mg single dose oral.
  Interventions: Drug: Nemonoxacin

INTERVENTIONS:
Drug: Nemonoxacin — Nemonoxacin Malate Capsules 500mg single dose oral
  Other Names: Nemonoxacin Malate Capsules

SUMMARY:
This is a single center, open-label, non-randomized, 1:1 parallel control and single dose administration study design. Healthy subjects will be matched to severe renal function impaired (eGFR≤30mL/min/1.73m2，CKD-EPI estimated) subjects in age, gender and weight as parallel control, which matches healthy with normal renal function according to the of subjects with impaired renal function as, after enrollment of subjects with severe impaired renal function (eGFR≤30mL/min/1.73m2，CKD-EPI estimated). Renal function impaired group and control group both receive orally single-dose of nemonoxacin malate capsule (0.5g). Collect the blood and urine samples before and after the administration to perform pharmacokinetic analysis and safety observation.

DETAILED DESCRIPTION:
Single dose study: evaluate safety and tolerability of oral nemonoxacin capsule 500mg

ELIGIBILITY:
Inclusion Criteria:

* Subjects with kidney impairment

  1. male or female aged 18 to 70 years；
  2. has a body mass index of 17 to 30 kg/m2;
  3. Patients with severe impaired renal function or end-stage renal disease (eGRF≤30ml/min/1.73m2, CKD-EPI estimated),and don't have hemodialysis.
  4. Female volunteers must meet:

     1. Has sterilization operation, or who are postmenopausal must have been postmenopausal for >1 year, or
     2. Has childbearing potential, but meet the requirement as following:

     Negative pregnancy test prior to enrollment, and Agree with use 1 medical accepted methods of birth control (eg. Hormonal contraceptive, barrier contraceptive with additional spermicide, or an intrauterine device) during the whole study and continuing until 1 month after the end of the study, and Non-breastfeeding;
  5. Male volunteers must agree to use medical accepted method of birth control (e.g. barrier contraceptive or sexual partner use the method as (4) above) during the study and through 1month after the end of study；
  6. Agree stay in ward prior to dosing within 48h, and agree not to take coffee, tea, chocolate, alcohol, grapefruit juice, orange juice and other food and drink which contain caffeine and xanthine；
  7. Can sign informed consent form on his own accord；
  8. Can comply with study procedures.
* Healthy subjects without renal impairment

  1. Male or female volunteers (matched to a subject with renal impairment in gender）；
  2. Aged 18 to 70 years (matched to a subject with renal impairment±5 years, matched range cannot exceed±5 years)；
  3. Has a body mass index of 17 to 30 kg/m2（matched to a subject with hepatic impairment±15%，matched range cannot exceed±15%）；
  4. Must be in good health as determined by screening medical history, physical examination, vital signs, laboratory test, B ultrasonography and chest X ray；
  5. Renal function is normal (eGFR≥90mL/min/1.73m2)
  6. Female volunteers must meet:

     1. Has sterilization operation, or who are postmenopausal must have been postmenopausal for >1 year, or
     2. Has childbearing potential, but meet the requirement as following:

     Negative pregnancy test prior to enrollment, and Agree with use 1 medical accepted methods of birth control (eg. Hormonal contraceptive, barrier contraceptive with additional spermicide, or an intrauterine device) during the whole study and continuing until 1 month after the end of the study, and Non-breastfeeding;
  7. Male volunteers must agree to use medical accepted method of birth control (e.g. barrier contraceptive or sexual partner use the method as (6) above) during the study and through 1month after the end of study；
  8. Agree stay in ward prior to dosing within 48h, and agree not to take coffee, tea,chocolate, alcohol, grapefruit juice, orange juice and other food and drink which contain caffeine and xanthine；
  9. Can sign informed consent form on his own accord；
  10. Can comply with study procedures

Exclusion Criteria:

* Subjects with kidney impairment

  1. Has known or suspected allergies to quinolones, fluoroquinolones,Nemonoxacin or excipients or allergic constitution；
  2. Has diseases (e.g. unstable cardiac disease, uncontrolled hypertension, uncontrolled asthma, uncontrolled diabetes, uncontrolled thyroid disease, uncontrolled epilepsy, myasthenia gravis or other neuromuscular disease, which may affect PK profile of drug in vivo or increase the risk in study except the disease caused renal function impaired;
  3. Has moderate or severe anemia (Hb<60g/L), severe hypertension (SBP>180mmHg and/or DBP>110mmHg) or diabetic nephropathy;
  4. Has history of clinically significant cardiovascular, neurological or psychiatric, gastrointestinal, pulmonary, renal, endocrine disease prior to study within 1 year；
  5. Has disease seriously affect the immune system such as hematological disease, malignant tumor, or taking immunosuppressant；
  6. Scr changes exceed more than 30% compared with baseline (Renal function tests two weeks before screening period ,even not conducted in this study can performed as baseline);
  7. Has uracratia or anuria;
  8. Has significant drug change including prescription drugs, non-prescription drugs or nutritional regimen 2 weeks before dosing(judged by investigator);
  9. Has administration of drug which eliminated mainly via kidney or damage kidney 2 weeks before dosing or need combination use in the study (e.g. TMP-SMZ or non-steroid anti-inflammatory drug);
  10. Has a history of alcoholism within 2 years prior to dosing; drink≥12 times within 3 months prior dosing; alcohol test positive as screening；
  11. Has history of drug misuse within 2 years prior to dosing; urine drug screen positive；
  12. Has history of taking products of tobacco or nicotine more than 5 cigarettes/day within 1 month prior to dosing, or cannot stop smoking during the study;
  13. Use of another investigational drug or drug which can damage hepatic function within 3 months prior to dosing；
  14. Has history of blood donation 3 months before study;
  15. Use of drugs affect function of liver metabolism enzyme (e.g. benzene, isopropyl amine, the barbiturates benzodiazepines, marijuana, cocaine, opiates and phencyclidine) within 30 days prior to dosing；
  16. Has to take the drug which may affect the PK profile of investigate drug (e.g. antacids, sucralfate, metal cation, calcium supplements, warfarin, nonsteroidal anti-inflammatory drugs, theophylline, cyclosporine, probenecid and cimetidine)；
  17. Has gastrointestinal disease or malabsorption syndrome affecting drug Absorb；
  18. Has history of seizures or central nervous system disease which the investigator considers to interfere with compliancy of protocol; or has risk of suicide；
  19. Clinical significant abnormal 12-lead electrocardiograms (ECGs) at screening (eg. atrioventricular block, torsades de pointes ventricular tachycardia (TdT), and other types of ventricular tachycardia, ventricular fibrillation, ventricular flutter, T wave change with clinical significance or any abnormal results of 12-lead ECG which affect QTc interphase)；
  20. HIVAb, HBsAg, HCVAb or syphilis RPR test positive;
  21. Not agree stay in ward prior to dosing within 48h, and agree not to take coffee, tea,chocolate, alcohol, grapefruit juice, orange juice and other food and drink which contain caffeine and xanthine；
  22. Conditions investigator consider not suitable to be enrolled in the study.
* Healthy subjects without kidney impairment

  1. Has known or suspected allergies to quinolones, fluoroquinolones, nemonoxacin or excipients or allergic constitution；
  2. Has a history of alcoholism within 2 years prior to dosing; drink≥12 times within 3 months prior dosing; alcohol test positive as screening；
  3. Has history of drug misuse within 2 years prior to dosing; urine drug screen positive；
  4. Has history of taking products of tobacco or nicotine more than 5 cigarettes/ day within 1 month prior to dosing, or cannot stop smoking during the study；
  5. Donated blood or use of another investigational drug within 3 months prior to dosing；
  6. Has history of chronic liver, renal, cardiovascular, neurological or psychiatric, gastrointestinal, pulmonary, urinary, endocrine disease cannot controlled by drugs；
  7. Use of drugs affect function of liver metabolism enzyme within 30 days prior to dosing; or need to take medications which may affect the PK profile of investigational drug (including: products containing Calcium, aluminum, magnesium, iron and zinc, sucralfate, antacid, nutrition supplements, Vitamins and metal supplements) during the study；
  8. Is taking any antibacterial agents；
  9. HIV-Ab, HBsAg ,HCV-Ab or syphilis RPR positive；
  10. Clinical significant abnormal 12-lead electrocardiograms (ECGs) at screening (eg. atrioventricular block, torsades de pointes ventricular tachycardia (TdT), and other types of ventricular tachycardia, ventricular fibrillation, ventricular flutter, T wave change with clinical significance or QTc>450ms) ；
  11. Has abnormal result of laboratory test with clinical significance assessed by investigator at screening；
  12. Has gastrointestinal disease or malabsorption syndrome affecting drug Absorb；
  13. Has history of seizures or central nervous system disease which the investigator considers to interfere with compliancy of protocol; or has risk of suicide；
  14. Has any antibacterials, glucocorticoids, immunosuppressive agents or drug may damage organs within 14 days prior to dosing；
  15. Cannot orally take drug；
  16. Has history of or currently has disease and condition may affect the safety and efficancy assessment of investigational drug judged by investigator；
  17. Conditions investigator consider not suitable to be enrolled in the study;
  18. Is a member of the clinical site personnel directly affiliated with this study；

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2017-04-05 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) parameters of single oral dose of nemonoxacin in severe impaired renal Function:maximum plasma drug concentration ( Cmax) | Pre-dose, 0.5h,1h, 1.5h, 2h, 4h, 6h, 8h, 12h, 24h, 48h, 72h after dosing
Pharmacokinetics (PK) parameters of single oral dose of nemonoxacin in severe impaired renal Function: time at which maximum plasma concentration is observed (Tmax) | Pre-dose, 0.5h,1h, 1.5h, 2h, 4h, 6h, 8h, 12h, 24h, 48h, 72h after dosing
Pharmacokinetics (PK) parameters of single oral dose of nemonoxacin in severe impaired renal Function: area under the plasma concentration vs. time curve (AUC0-t and AUC0-∞) | Pre-dose, 0.5h,1h, 1.5h, 2h, 4h, 6h, 8h, 12h, 24h, 48h, 72h after dosing
Pharmacokinetics (PK) parameters of single oral dose of nemonoxacin in severe impaired renal Function: elimination half-life (t1/2) | Pre-dose, 0.5h,1h, 1.5h, 2h, 4h, 6h, 8h, 12h, 24h, 48h, 72h after dosing
Pharmacokinetics (PK) parameters of single oral dose of nemonoxacin in severe impaired renal Function: mean dissolution time(MRT) | Pre-dose, 0.5h,1h, 1.5h, 2h, 4h, 6h, 8h, 12h, 24h, 48h, 72h after dosing
Pharmacokinetics (PK) parameters of single oral dose of nemonoxacin in severe impaired renal Function: total clearance of the drug from plasma (CLz/F) | Pre-dose, 0.5h,1h, 1.5h, 2h, 4h, 6h, 8h, 12h, 24h, 48h, 72h after dosing
Pharmacokinetics (PK) parameters of single oral dose of nemonoxacin in severe impaired renal Function: Apparent Volume of Distribution (Vz/F) | Pre-dose, 0.5h,1h, 1.5h, 2h, 4h, 6h, 8h, 12h, 24h, 48h, 72h after dosing
Pharmacokinetics (PK) parameters of single oral dose of nemonoxacin in severe impaired renal Function: cumulative amount of unchanged drug excreted into the urine (Ae Urine 0-24h,0-72h） | Within 72h after dosing
Pharmacokinetics (PK) parameters of single oral dose of nemonoxacin in severe impaired renal Function::renal clearance of the drug from plasma (CLr) | Within 72h after dosing
Pharmacokinetics (PK) parameters of single oral dose of nemonoxacin in severe impaired renal Function:minimum plasma drug concentration (Cmin) | Pre-dose, 0.5h,1h, 1.5h, 2h, 4h, 6h, 8h, 12h, 24h, 48h, 72h after dosing]

SECONDARY OUTCOMES:
Safety assessed by AEs | up to 72 hours after study drug dosing
  reported spontaneously or not by leading questions
Safety assessed by vital signs-respiratory rate | up to 72 hours after study drug dosing
  respiratory rate, "times per minute"
Safety assessed by vital signs-body temperature | up to 72 hours after study drug dosing
  body temperature, "degree centigrade"
Safety assessed by vital signs-blood pressure | up to 72 hours after study drug dosing
  blood pressure, "mmHg"
Safety assessed by vital signs-pulse rate | up to 72 hours after study drug dosing
  pulse rate, "beats per minute"
Number of Participants with Abnormal Laboratory Values | up to 72 hours after study drug dosing
  Hematology, blood biochemistry,cogulation test and urinalysis
Safety assessed by physical examination | up to 72 hours after study drug dosing
  (1) general appearance (2) skin (3) head and neck (4)chest, including heart, pulmonary and breast (5) abdomen, including stomach and intestines, liver and gallbladder (6) back (7) Urinary tract (8) extremity (9) neurological or psychiatric system (10) lymph gland (11)others.
Safety assessed by 12-lead ECGs | up to 72 hours after study drug dosing

CONTACTS AND LOCATIONS:
Locations (1):
- ZheJiang Medicine, Shaoxing, China

IPD SHARING:
Plan to Share IPD: Yes